CLINICAL TRIAL: NCT04339231
Title: Block of the Sphenopalatine Nerve Ganglion for Postoperative Analgesia in Transsphenoidal Approaches: a Prospective, Randomized and Double-blind Study
Brief Title: Block of the Sphenopalatine Nerve Ganglion for Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Alexandra Rezende Assad, PhD, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sphenopalatine
Record Dates: First submitted 2020-03-31; First posted 2020-04-09 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Surgery; Anesthesia, Local; Postoperative Pain
Keywords: ropivacaine; sphenopalatine
MeSH Terms: conditions — Pain, Postoperative | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: XXXXX
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine group (Active Comparator): The block of the sphenopalatine ganglion will be performed bilaterally through a cotton bud soaked with the anesthetic solution ropivacaine, at a concentration of 1%, advancing it through the nasal cavities towards the posterior nasopharynx wall. A slight resistance in the progression of the cottonoid indicates its contact with the mucosa of the posterior pharyngeal wall. The cottonoid will remain in this position for 20 minutes, so that there is absorption of the anesthetic solution through the mucosa up to the sphenopalatine ganglion, which, in general, is found anatomically around 3 millimeters in depth from the surface. After the established time, the cotton buds are removed.
  Interventions: Procedure: sphenopalatine ganglion block
- Saline 0,9% group (Placebo Comparator): The block of the sphenopalatine ganglion will be performed bilaterally through a cotton bud soaked with saline solution, in a concentration of 0.9%, advancing it through the nasal cavities towards the posterior wall of the nasopharynx. A slight resistance in the progression of the cottonoid indicates its contact with the mucosa of the posterior pharyngeal wall. The cottonoid will remain in this position for 20 minutes, so that the solution is absorbed by the mucosa up to the sphenopalatine ganglion, which, in general, is anatomically three millimeters deep from the surface. After the established time, the cotton buds are removed.
  Interventions: Procedure: sphenopalatine ganglion block

INTERVENTIONS:
Procedure: sphenopalatine ganglion block — The block of the sphenopalatine ganglion will be performed bilaterally, using a cotton bud soaked with 1% ropivacaine, placed in the mucosa of the posterior wall of the nasal cavity, through both nostrils.
  Once placed in the proper position, the swab will remain for about 20 minutes to absorb the local anesthetic from the mucosa.

SUMMARY:
Transsphenoidal surgery is considered safe and effective and is currently the procedure of choice for the removal of intrasellar lesions. Direct transnasal access to the sphenoid sinus, without the need for detachment of the nasal septum, provides less postoperative morbidity compared to traditional methods. Sphenopalatine ganglion block is known for its efficacy in otorhinolaryngological surgeries in which the sinuses are approached by transnasal endoscopy, as an important part of postoperative analgesia. However, in a neurosurgical environment, specifically in the treatment of tumors of the sella turcica, the use of the blockade of the referred ganglion to produce postoperative analgesia has been used in a scarce way in the literature. The primary objective of the study is to verify whether blocking the sphenopalatine nerve ganglion in the nasopharynx posterior wall provides better postoperative pain control in surgeries with nasal access for transsphenoidal approach, compared to the placebo group. As secondary objectives, the investigators will observe the consumption of opioids in the intraoperative period, in addition to the incidence of nausea, vomiting and postoperative headache also within 24 hours. Forty patients with physical status P1, P2 or P3 will be prospectively analyzed by the American Society of Anesthesiology (ASA) to undergo microsurgery for tumors with a sellar and / or suprasellar location, with transsphenoidal access, in patients with an age range between 18 and 64 years old, including men and women.

DETAILED DESCRIPTION:
Transsphenoidal surgery is considered safe and effective and is currently the procedure of choice for the removal of intrasellar lesions. Direct transnasal access to the sphenoid sinus, without the need for detachment of the nasal septum, provides less postoperative morbidity compared to traditional methods. Sphenopalatine ganglion block is known for its efficacy in otorhinolaryngological surgeries in which the sinuses are approached by transnasal endoscopy, as an important part of postoperative analgesia. However, in a neurosurgical environment, specifically in the treatment of tumors of the sella turcica, the use of the blockade of the referred ganglion to produce postoperative analgesia has been used in a scarce way in the literature. The primary objective of the study is to verify whether blocking the sphenopalatine nerve ganglion in the nasopharynx posterior wall provides better postoperative pain control in surgeries with nasal access for transsphenoidal approach, compared to the placebo group. As secondary objectives, the investigators will observe the consumption of opioids in the intraoperative period, in addition to the incidence of nausea, vomiting and postoperative headache also within 24 hours. Forty patients with physical status P1, P2 or P3 will be prospectively analyzed by the American Society of Anesthesiology (ASA) to undergo microsurgery for tumors with a sellar and / or suprasellar location, with transsphenoidal access, in patients with an age range between 18 and 64 years old, including men and women. As for the surgical technique, both the use of the microscope and the endoscope will be considered. They will be randomly allocated to a placebo group (group P; 0.9% saline, n = 20) and a test group (group R; ropivacaine 1%, n = 20).

ELIGIBILITY:
Inclusion Criteria:

1. Both genders;
2. Age between 18 and 64 years;
3. Physical status according to the American Society of Anesthesiologists (ASA) I, II and III
4. Saddle or suprasellar tumors with transsphenoidal access;

Exclusion Criteria:

1. Participation in another study in the last month;
2. Patients with a history of chronic pain;
3. Previous surgeries with a transsphenoidal approach;
4. Known hypersensitivity to ropivacaine;
5. Patient's refusal;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-25 (Estimated); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-04-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative analgesia using the visual analogue pain scale (VAS pain) | Immediately after awakening from anesthesia
  To verify whether blocking the sphenopalatine nerve ganglion in the posterior nasopharynx wall provides change in postoperative pain control, assessed using the visual analogue pain scale, in surgeries with nasal access for transsphenoidal approach, compared to the placebo group.
Evaluation of postoperative analgesia using the visual analogue pain scale (VAS pain) | 2 hours postoperative
  To verify whether blocking the sphenopalatine nerve ganglion in the posterior nasopharynx wall provides change in postoperative pain control, assessed using the visual analogue pain scale, in surgeries with nasal access for transsphenoidal approach, compared to the placebo group.
Evaluation of postoperative analgesia using the visual analogue pain scale (VAS pain) | 6 hours postoperative
  To verify whether blocking the sphenopalatine nerve ganglion in the posterior nasopharynx wall provides change in postoperative pain control, assessed using the visual analogue pain scale, in surgeries with nasal access for transsphenoidal approach, compared to the placebo group.
Evaluation of postoperative analgesia using the visual analogue pain scale (VAS pain) | 12 hours postoperative
  To verify whether blocking the sphenopalatine nerve ganglion in the posterior nasopharynx wall provides change in postoperative pain control, assessed using the visual analogue pain scale, in surgeries with nasal access for transsphenoidal approach, compared to the placebo group.
Evaluation of postoperative analgesia using the visual analogue pain scale (VAS pain) | 24 hours postoperative
  To verify whether blocking the sphenopalatine nerve ganglion in the posterior nasopharynx wall provides change in postoperative pain control, assessed using the visual analogue pain scale, in surgeries with nasal access for transsphenoidal approach, compared to the placebo group.

SECONDARY OUTCOMES:
Change the consumption of intraoperative opioids | Intraoperative time
  Check the change in total opioid consumption in the intraoperative period
Use of complementary opioids | Immediately after awakening from anesthesia
  Assess the number of rescue doses with opioids in pos operative period for for adequate analgesia (it is understood as insufficient analgesia classification on the visual analog scale of pain greater than or equal to 3)
Use of complementary opioids | 2 hours postoperative
  Assess the number of rescue doses with opioids in pos operative period for for adequate analgesia (it is understood as insufficient analgesia classification on the visual analog scale of pain greater than or equal to 3)
Use of complementary opioids | 6 hours postoperative
  Assess the number of rescue doses with opioids in pos operative period for for adequate analgesia (it is understood as insufficient analgesia classification on the visual analog scale of pain greater than or equal to 3)
Use of complementary opioids | 12 hours postoperative
  Assess the number of rescue doses with opioids in pos operative period for for adequate analgesia (it is understood as insufficient analgesia classification on the visual analog scale of pain greater than or equal to 3)
Use of complementary opioids | 24 hours postoperative
  Assess the number of rescue doses with opioids in pos operative period for for adequate analgesia (it is understood as insufficient analgesia classification on the visual analog scale of pain greater than or equal to 3)
Postoperative nausea and vomiting; | Immediately after awakening from anesthesia
  Check the incidence of postoperative nausea and vomiting
Postoperative nausea and vomiting; | 2 hours postoperative
  Check the incidence of postoperative nausea and vomiting
Postoperative nausea and vomiting; | 6 hours postoperative
  Check the incidence of postoperative nausea and vomiting
Postoperative nausea and vomiting; | 12 hours postoperative
  Check the incidence of postoperative nausea and vomiting
Postoperative nausea and vomiting; | 24 hours postoperative
  Check the incidence of postoperative nausea and vomiting
Postoperative headache | Immediately after awakening from anesthesia
  Check the incidence of postoperative headache
Postoperative headache | 2 hours postoperative
  Check the incidence of postoperative headache
Postoperative headache | 6 hours postoperative
  Check the incidence of postoperative headache
Postoperative headache | 12 hours postoperative
  Check the incidence of postoperative headache
Postoperative headache | 24 hours postoperative
  Check the incidence of postoperative headache

CONTACTS AND LOCATIONS:
Overall Officials: Ismar S Cavalcanti, MD., Study Chair — Universidade Federal Fluminense
Locations (1):
- Instituto Estadual do Cérebro Paulo Niemeyer, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual patient data

REFERENCES:
- [Result] Liu JK, Das K, Weiss MH, Laws ER Jr, Couldwell WT. The history and evolution of transsphenoidal surgery. J Neurosurg. 2001 Dec;95(6):1083-96. doi: 10.3171/jns.2001.95.6.1083. PMID 11765830
- [Result] Kesimci E, Ozturk L, Bercin S, Kiris M, Eldem A, Kanbak O. Role of sphenopalatine ganglion block for postoperative analgesia after functional endoscopic sinus surgery. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):165-9. doi: 10.1007/s00405-011-1702-z. Epub 2011 Jul 8. PMID 21739090
- [Result] Cho DY, Drover DR, Nekhendzy V, Butwick AJ, Collins J, Hwang PH. The effectiveness of preemptive sphenopalatine ganglion block on postoperative pain and functional outcomes after functional endoscopic sinus surgery. Int Forum Allergy Rhinol. 2011 May-Jun;1(3):212-8. doi: 10.1002/alr.20040. Epub 2011 Apr 13. PMID 22287376
- See also: Endoscopic transnasal approach to sellar tumors — http://www.scielo.br/scielo.php?pid=S0034-72992007000400005&script=sci_abstract&tlng=pt
- See also: Sphenopalatine ganglion block for postdural puncture headache in ambulatory setting — http://www.scielo.br/pdf/rba/v67n3/0034-7094-rba-67-03-0311.pdf
- See also: Role of Intraoperative Endoscopic Sphenopalatine Ganglion Block in Sinonasal Surgery — http://scialert.net/fulltext/?doi=jms.2007.1297.1303

DOCUMENTS (1):
  • Informed Consent Form (2019-11-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT04339231/ICF_000.pdf